CLINICAL TRIAL: NCT07324213
Title: Evaluation of the Degree of Regeneration of Post-Extraction Alveolar Sockets of Mandibular Third Molars Using Tissue Engineering and Photobiomodulation
Brief Title: Healing of Mandibular Third Molar Extraction Sockets Using Platelet Concentrates and Photobiomodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Innovation Center Wroclaw (Other)
Collaborators: Wrocław Medical University (Unknown)
Responsible Party: Principal Investigator, Jakub Hadzik, Associate Professor, PhD, DSc (Med.), Specialist in Oral Surgery, Medical Innovation Center Wroclaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB7052019-UMW
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Impacted Mandibular Third Molar; Alveolar Bone Loss; Impacted Mandibular Third Molar Extraction
Keywords: Mandibular third molar extraction,; Platelet-rich fibrin,; Concentrated growth factors,; Fractal dimension analysis; Low-level laser therapy,; Photobiomodulation,; Bone regeneration,
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of six parallel intervention groups and received only the intervention allocated to their study arm.
Who Masked: Participant
Masking Description: Participants were not informed about the type of regenerative intervention applied. Due to the nature of the surgical procedures, care providers and investigators were not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control - Standard Extraction (Other): Participants underwent surgical extraction of an impacted mandibular third molar followed by standard primary wound closure without the use of platelet concentrates or photobiomodulation.
  Interventions: Procedure: Mandibular Third Molar Extraction With Primary Wound Closure
- Photobiomodulation (Other): Participants underwent surgical extraction of an impacted mandibular third molar followed by primary wound closure and photobiomodulation using low-level laser therapy applied immediately after surgery and during follow-up visits.
  Interventions: Procedure: Mandibular Third Molar Extraction With Primary Wound Closure; Other: Photobiomodulation
- A-PRF+ (Other): Participants underwent surgical extraction of an impacted mandibular third molar followed by placement of autologous advanced platelet-rich fibrin (A-PRF+) into the extraction socket prior to primary wound closure.
  Interventions: Procedure: Mandibular Third Molar Extraction With Primary Wound Closure; Biological: Autologous Platelet Concentrates
- CGF (Other): Participants underwent surgical extraction of an impacted mandibular third molar followed by placement of autologous concentrated growth factors (CGF) into the extraction socket prior to primary wound closure.
  Interventions: Procedure: Mandibular Third Molar Extraction With Primary Wound Closure; Biological: Autologous Platelet Concentrates
- A-PRF+ Plus Photobiomodulation (Other): Participants underwent surgical extraction of an impacted mandibular third molar followed by placement of autologous advanced platelet-rich fibrin (A-PRF+) into the extraction socket and adjunctive photobiomodulation using low-level laser therapy.
  Interventions: Procedure: Mandibular Third Molar Extraction With Primary Wound Closure; Biological: Autologous Platelet Concentrates; Other: Photobiomodulation
- CGF Plus Photobiomodulation (Other): Participants underwent surgical extraction of an impacted mandibular third molar followed by placement of autologous concentrated growth factors (CGF) into the extraction socket and adjunctive photobiomodulation using low-level laser therapy.
  Interventions: Procedure: Mandibular Third Molar Extraction With Primary Wound Closure; Biological: Autologous Platelet Concentrates; Other: Photobiomodulation

INTERVENTIONS:
Procedure: Mandibular Third Molar Extraction With Primary Wound Closure — Surgical extraction of a partially or fully impacted mandibular third molar performed under standardized clinical conditions, followed by primary wound closure with sutures. This procedure was applied in all study arms.
Biological: Autologous Platelet Concentrates — Autologous platelet concentrates prepared from the participant's peripheral blood and placed into the extraction socket prior to primary wound closure. Advanced platelet-rich fibrin (A-PRF+) and concentrated growth factors (CGF) were obtained using standardized centrifugation protocols and used according to the allocated study arm.
  Other Names: Advanced Platelet-Rich Fibrin (A-PRF+); Concentrated Growth Factors (CGF)
  Arms: A-PRF+; A-PRF+ Plus Photobiomodulation; CGF; CGF Plus Photobiomodulation
Other: Photobiomodulation — Adjunctive photobiomodulation performed using low-level laser therapy applied to the extraction site. The intervention was delivered immediately after surgery and during follow-up visits according to the study protocol.
  Arms: A-PRF+ Plus Photobiomodulation; CGF Plus Photobiomodulation; Photobiomodulation

SUMMARY:
Surgical removal of impacted mandibular third molars is a common procedure that may be associated with postoperative pain, swelling, limited mouth opening, and delayed bone healing. Various regenerative techniques are used to improve healing outcomes after tooth extraction.

This study evaluated whether autologous platelet concentrates (advanced platelet-rich fibrin [A-PRF+] and concentrated growth factors [CGF]) and photobiomodulation using low-level laser therapy can improve healing after mandibular third molar extraction.

Participants requiring surgical removal of a mandibular third molar were randomly assigned to one of six treatment groups. Depending on the group, patients received standard wound closure alone, photobiomodulation, placement of autologous platelet concentrates into the extraction socket, or a combination of platelet concentrates and photobiomodulation.

Postoperative pain, swelling, mouth opening, and early wound healing were assessed during the first postoperative week. Bone regeneration within the extraction socket was evaluated using radiological imaging several months after surgery.

All procedures used in this study are commonly applied in clinical practice and are considered safe. The results of this study may help identify the most effective approach to improve healing and reduce postoperative discomfort following mandibular third molar extraction.

DETAILED DESCRIPTION:
Surgical extraction of impacted mandibular third molars frequently results in postoperative complications such as pain, edema, trismus, and delayed bone regeneration. Advances in regenerative medicine have introduced autologous platelet concentrates, including advanced platelet-rich fibrin (A-PRF+) and concentrated growth factors (CGF), which provide sustained release of growth factors that may enhance soft and hard tissue healing. Additionally, photobiomodulation using low-level laser therapy has been reported to reduce inflammation and stimulate tissue regeneration.

This single-center, randomized, single-blind clinical trial was conducted to evaluate the effectiveness of A-PRF+, CGF, and photobiomodulation, applied alone or in combination, in enhancing postoperative healing following mandibular third molar extraction.

A total of 122 generally healthy adult participants requiring surgical extraction of a partially or fully impacted mandibular third molar were enrolled. Participants were randomly allocated to one of six parallel study groups: standard extraction with primary wound closure (control), extraction with photobiomodulation, extraction with socket augmentation using A-PRF+, extraction with socket augmentation using CGF, extraction with A-PRF+ combined with photobiomodulation, or extraction with CGF combined with photobiomodulation. All surgical procedures were performed under standardized clinical conditions. Primary wound closure was attempted in all cases. Photobiomodulation was performed using a diode laser with a wavelength of 635 nm, power output of 100 mW, and energy density of 4 J/cm², applied at four points around the extraction socket. Autologous platelet concentrates were prepared from the patient's peripheral blood using standardized centrifugation protocols.

Clinical outcomes, including postoperative pain assessed using a visual analogue scale, facial swelling, mouth opening, and early wound healing, were evaluated at 1, 3, and 7 days after surgery. Radiological assessment of bone regeneration within the extraction socket was performed 3 to 4 months postoperatively using cone-beam computed tomography-based fractal dimension analysis.

The study was conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines. All participants provided written informed consent prior to enrollment. The findings of this study aim to contribute to the optimization of postoperative management following mandibular third molar extraction by identifying effective regenerative treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 40 years.
* Indication for surgical extraction of a partially or fully impacted mandibular third molar.
* Generally healthy individuals without systemic diseases.
* Ability to provide written informed consent.
* Willingness to attend scheduled follow-up visits.

Exclusion Criteria:

* Presence of systemic diseases or metabolic disorders.
* Pregnancy or breastfeeding.
* Smoking.
* Recent antibiotic therapy.
* Poor oral hygiene.
* Exceptionally difficult tooth position.
* Surgical procedure exceeding the expected duration.
* Inability to achieve primary wound closure.
* Failure to comply with follow-up visits.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | 1 day, 3 days, and 7 days after surgery
  Postoperative pain intensity was assessed using a visual analogue scale (VAS) ranging from 1 to 10, where 1 indicates no pain and 10 indicates the worst pain imaginable.
Alveolar Bone Regeneration | 4 months after surgery
  Bone regeneration within the post-extraction socket assessed using cone-beam computed tomography-based fractal dimension analysis.

SECONDARY OUTCOMES:
Postoperative Swelling | 1 day, 3 days, and 7 days after surgery
  Facial swelling assessed using standardized clinical measurements.
Postoperative Trismus | 1 day, 3 days, and 7 days after surgery
  Maximum mouth opening assessed by measuring interincisal distance.
Early Wound Healing | 7 days after surgery
  Early soft tissue healing was evaluated using the Early Healing Index (EHI), an ordinal scale with scores ranging from 1 (very poor soft tissue healing) to 5 (excellent soft tissue healing), with higher scores indicating a more favorable healing outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Medyczne Centrum Innowacji Wrocław Sp. z o.o., Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional data protection policies and the need to protect participant privacy. Aggregated and anonymized results are reported in publications arising from this study.